CLINICAL TRIAL: NCT01840228
Title: Vaginal Progesterone for the Prevention of Preterm Birth in Women With Arrested Preterm Labor
Acronym: PAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Washington University School of Medicine (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201301148
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-05

CONDITIONS: Premature Birth; Obstetric Labor, Premature
Keywords: Preterm; Progesterone
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Micronized progesterone suppository (Active Comparator): Micronized progesterone suppository 200 mg vaginally daily until 36 6/7 weeks' gestation.
  Interventions: Drug: Micronized progesterone suppository
- Placebo suppository (Placebo Comparator): One placebo suppository vaginally daily until 36 6/7 weeks' gestation.
  Interventions: Drug: Micronized progesterone suppository

INTERVENTIONS:
Drug: Micronized progesterone suppository

SUMMARY:
Preterm birth, defined as birth before 37 weeks' gestation, is a leading cause of infant death and disease. Progesterone is the single most effective intervention in the prevention of preterm birth. However, current use of this therapy is limited to certain high-risk groups including women with a history of preterm birth and women with a short cervix. This study seeks to evaluate the efficacy of this preventive therapy in another high-risk group: women with arrested preterm labor. The investigators hypothesize that administration of vaginal progesterone in women who present with preterm labor but remain undelivered 12 hours after cessation of short-term therapy to inhibit contractions will result in lower rates of preterm birth before 37 weeks' than will administration of placebo.

DETAILED DESCRIPTION:
RESEARCH DESIGN AND METHODS

The investigators will perform a randomized, blinded, placebo-controlled trial to evaluate the use of vaginal progesterone in women with arrested preterm labor after 24 weeks' gestation to reduce the risk of preterm birth before 37 weeks' gestation. Women enrolled in the study will be randomized to daily vaginal administration of progesterone (200 mg) or placebo from time of enrollment until 36 6/7 weeks' gestation. Women will be eligible if they have a singleton or twin gestation between 24 0/7 and 33 6/7 weeks' gestation and initially present with regular uterine contractions and a clinical diagnosis of preterm labor but remain undelivered without further cervical change 12 hours after discontinuation of acute tocolytic therapy. Women may also participate if it has been less than if they are considered eligible for discharge based on attending physician judgement prior to the 12 hour period of time.

Randomization and Blinding- Participants in the study will be randomized using a computer-generated randomization scheme with 1:1 allocation to receive progesterone or placebo. Investigators and research team members, participants, and the obstetric providers will be blinded to the allocated intervention.

Procedures-

* Data collection- Information will be recorded from the participant's medical record. Additional study information not included in the medical record will be obtained directly from the participant in an interview with the research team member.
* Follow-up- Regardless of whether the participant remains hospitalized or is discharged prior to delivery, she will meet with a study coordinator every 2 weeks. During the follow-up visit, a study team member will discuss compliance with the study drug and possible side effects. The participant will fill out a 1-page questionnaire that asks questions about compliance and side effects. This information will be recorded and provided to the Data Safety and Monitoring Board at the midpoint review.

SAMPLE SIZE ESTIMATION

The investigators plan to enroll 120 patients, with a 1:1 allocation to treatment and placebo. This sample size is adequate to detect a one-half reduction in the primary outcome, delivery before 37 weeks.

STATISTICAL ANALYSIS

Baseline characteristics of women randomized to progesterone will be compared with women randomized to placebo. Rates of delivery before 37 weeks' gestation will be compared among the groups using the Chi-square test. Secondary outcomes will be evaluated using the Chi-square test for binary outcomes and the Student t-test for continuous outcomes. Length of time from enrollment to delivery will be analyzed using Kaplan-Meier curves and the Cox proportional hazards model. All analyses will be performed using the intention-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Singleton or twin gestation
* Estimated gestational age between 24 0/7 and 33 6/7 weeks' gestation
* Initially present with regular contractions and clinical diagnosis of preterm labor but remain undelivered with 1) no further cervical change 12 hours after discontinuation of acute tocolytic therapy; or 2) be considered eligible for discharge based on attending physician judgment prior to the 12 hour period of time
* The participant's cervix must be at least 1 cm at the time of enrollment

Exclusion Criteria:

* Non-English speaking
* Rupture of membranes
* Chorioamnionitis
* Non-reassuring fetal status
* Maternal indication for delivery
* Placental abruption
* Intrauterine fetal demise
* Prenatally diagnosed major fetal anomaly
* Cervical cerclage in place
* Previous administration of progesterone during the current pregnancy for a history of preterm birth or short cervix
* Participant is either unwilling or unable to attend follow-up study visits following hospital discharge

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2018-05-07 (Actual); Study Completion 2018-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Macones, MD, MSCE, Study Chair — Washington University School of Medicine; Heather A Frey, MD, MSCI, Principal Investigator — Ohio State University
Locations (1):
- Washington University School of Medicine/ Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Background] Lyell DJ, Pullen KM, Mannan J, Chitkara U, Druzin ML, Caughey AB, El-Sayed YY. Maintenance nifedipine tocolysis compared with placebo: a randomized controlled trial. Obstet Gynecol. 2008 Dec;112(6):1221-1226. doi: 10.1097/AOG.0b013e31818d8386. PMID 19037029
- [Background] Likis FE, Edwards DR, Andrews JC, Woodworth AL, Jerome RN, Fonnesbeck CJ, McKoy JN, Hartmann KE. Progestogens for preterm birth prevention: a systematic review and meta-analysis. Obstet Gynecol. 2012 Oct;120(4):897-907. doi: 10.1097/AOG.0b013e3182699a15. PMID 22955308
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Fonseca EB, Celik E, Parra M, Singh M, Nicolaides KH; Fetal Medicine Foundation Second Trimester Screening Group. Progesterone and the risk of preterm birth among women with a short cervix. N Engl J Med. 2007 Aug 2;357(5):462-9. doi: 10.1056/NEJMoa067815. PMID 17671254
- [Background] Borna S, Sahabi N. Progesterone for maintenance tocolytic therapy after threatened preterm labour: a randomised controlled trial. Aust N Z J Obstet Gynaecol. 2008 Feb;48(1):58-63. doi: 10.1111/j.1479-828X.2007.00803.x. PMID 18275573
- [Background] Arikan I, Barut A, Harma M, Harma IM. Effect of progesterone as a tocolytic and in maintenance therapy during preterm labor. Gynecol Obstet Invest. 2011;72(4):269-73. doi: 10.1159/000328719. Epub 2011 Nov 12. PMID 22086108

RESULTS

PARTICIPANT FLOW:
Groups:
- Micronized Progesterone Suppository: Micronized progesterone suppository 200 mg vaginally daily until 36 6/7 weeks' gestation.
  Micronized progesterone suppository
- Placebo Suppository: One placebo suppository vaginally daily until 36 6/7 weeks' gestation.
  Micronized progesterone suppository
Period: Overall Study
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (5.5) | 26.3 (4.6) | 26.0 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 6 | 7 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38
Parity [Median (Inter-Quartile Range); unit: births] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 25.3 (7.9) | 25.4 (8.3) | 25.3 (8.0)
Prior preterm birth [Count of Participants; unit: Participants] | 6 | 8 | 14
Twin gestation [Count of Participants; unit: Participants] | 4 | 4 | 8
Marital status [Count of Participants; unit: Participants]
  Single | 13 | 11 | 24
  Married | 6 | 6 | 12
  Divorced | 0 | 1 | 1
  Unknown | 0 | 1 | 1
Insurance use [Count of Participants; unit: Participants]
  Public insurance | 14 | 11 | 25
  Private insurance | 3 | 7 | 10
  Other | 2 | 1 | 3
Gestational age at enrollment [Median (Inter-Quartile Range); unit: weeks] | 30.6 [29.9 to 32.9] | 30.4 [28.1 to 32.6] | 30.5 [29.3 to 32.6]
Cervical dilation at admission [Median (Inter-Quartile Range); unit: cm] | 1.5 [1 to 3] | 1 [1 to 2] | 1.25 [1 to 3]
Cervical dilation at enrollment [Median (Inter-Quartile Range); unit: cm] | 3 [1.5 to 4] | 2.5 [1 to 3] | 2.75 [1.5 to 3]
Tobacco use [Count of Participants; unit: Participants] | 3 | 4 | 7
Prior use of progesterone (17OHP-C) [Count of Participants; unit: Participants] | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Delivered Before 37 Weeks'
Time Frame: Duration of current pregnancy, anticipated maximum 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Number analyzed (Participants) | 18 | 18
Participants | 11 | 10
Statistical Analysis 1: Comparison: Micronized Progesterone Suppository vs Placebo Suppository; Test type: Superiority; p = 0.74, Chi-squared; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.63 to 1.91]

2. Secondary Outcome: Number of Participants Who Delivered Before 34 Weeks'
Description: Evaluated in women enrolled prior to 32 weeks gestation
Time Frame: Duration of current pregnancy, anticipated maximum 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Number analyzed (Participants) | 14 | 12
Participants | 3 | 6
Statistical Analysis 1: Comparison: Micronized Progesterone Suppository vs Placebo Suppository; Test type: Superiority; p = 0.13, Fisher Exact; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.14 to 1.36]

3. Secondary Outcome: Delivery Within 2 Weeks of Randomization
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Number analyzed (Participants) | 18 | 18
Participants | 6 | 4
Statistical Analysis 1: Comparison: Micronized Progesterone Suppository vs Placebo Suppository; Test type: Superiority; p = 0.71, Fisher Exact; Risk Ratio (RR) = 1.50, 95% CI 2-sided [0.51 to 4.43]

4. Secondary Outcome: Number of Weeks Pregnancy Prolongation
Time Frame: Duration of current pregnancy, anticipated maximum 18 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Number analyzed (Participants) | 18 | 18
weeks | 5.3 [1.3 to 6.7] | 5.0 [2.0 to 8.0]
Statistical Analysis 1: Comparison: Micronized Progesterone Suppository vs Placebo Suppository; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Infant Birth Weight
Time Frame: Day of delivery in current pregnancy
Measure: Mean (Standard Deviation); unit: grams
Groups:
- Micronized Progesterone Suppository - SINGLETON: Micronized progesterone suppository 200 mg vaginally daily until 36 6/7 weeks' gestation in singleton subgroup.
  Micronized progesterone suppository
- Placebo Suppository - SINGLETON: One placebo suppository vaginally daily until 36 6/7 weeks' gestation in singleton subgroup
  Micronized progesterone suppository
- Micronized Progesterone Suppository - TWINS: Micronized progesterone suppository 200 mg vaginally daily until 36 6/7 weeks' gestation in twin subgroup.
  Micronized progesterone suppository
- Placebo Suppository - TWINS: One placebo suppository vaginally daily until 36 6/7 weeks' gestation in twin subgroup
  Micronized progesterone suppository
Arm/Group | Micronized Progesterone Suppository - SINGLETON | Placebo Suppository - SINGLETON | Micronized Progesterone Suppository - TWINS | Placebo Suppository - TWINS
Number analyzed (Participants) | 14 | 14 | 8 | 8
grams | 2454.9 (659.4) | 2523.1 (748.5) | 2164.4 (215.9) | 1974.1 (252.8)

6. Secondary Outcome: Neonatal Intensive Care Unit Admission
Time Frame: Followed for duration of neonatal hospital stay, estimated maximum 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository - SINGLETON | Placebo Suppository - SINGLETON | Micronized Progesterone Suppository - TWINS | Placebo Suppository - TWINS
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants | 2 | 2 | 0 | 1

7. Secondary Outcome: Number of Participants With Chorioamnionitis
Time Frame: Duration of current pregnancy, anticipated maximum 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

8. Secondary Outcome: Composite Neonatal Outcome
Description: A composite neonatal outcome comprising neonatal death, respiratory distress syndrome, bronchopulmonary dysplasia, severe (grade III/IV) interventricular hemorrhage, necrotizing enterocolitis, and sepsis.
Time Frame: Followed for duration of neonatal hospital stay, estimated maximum 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Micronized Progesterone Suppository - SINGLETON | Placebo Suppository - SINGLETON | Micronized Progesterone Suppository - TWINS | Placebo Suppository - TWINS
Number analyzed (Participants) | 14 | 14 | 8 | 8
Participants | 5 | 5 | 3 | 7

ADVERSE EVENTS:
Time Frame: Information about adverse events was collected from time of enrollment until discharge from the hospital after delivery for all participants, which is generally < 1 week after delivery
Arm/Group | Micronized Progesterone Suppository | Placebo Suppository
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Micronized Progesterone Suppository (N=18) | Placebo Suppository (N=18)
Vaginal discharge (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Vaginal irritation (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Other (General disorders) | 0 (0) | 3 (3) — Includes swelling of extremities, dizziness and fatigue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT01840228/Prot_SAP_000.pdf